CLINICAL TRIAL: NCT01648725
Title: Influence of Hypnosis on the Propofol Requirement to Induce General Anesthesia
Brief Title: Hypnosis and Closed-Loop Anesthesia System
Acronym: LoopHypnosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/12; 2012-A00369-34 (Other: AFSSAPS)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia
Keywords: Hypnosis; Anesthesia; Propofol; Closed-loop
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis (Experimental): standard care plus hypnosis followed by closed-loop administration of propofol for anesthesia induction
  Interventions: Procedure: Hypnosis
- Control (Active Comparator): standard care without hypnosis followed by closed-loop administration of propofol for anesthesia induction
  Interventions: Procedure: usual care

INTERVENTIONS:
Procedure: Hypnosis — A short preanesthetic hypnosis before induction of anesthesia
  Arms: Hypnosis
Procedure: usual care — Standard care before induction of anesthesia
  Arms: Control

SUMMARY:
Hypnosis may reduce patient anxiety. The main goal of this study is to determine in what extent, hypnosis decreases propofol requirement to induce induction of general anesthesia.

A particular aspect of this study is that induction is provided by a closed-loop system which delivers propofol according to bispectral index.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for a surgical procedure under general anesthesia

Exclusion Criteria:

* pregnancy, breast feeding woman
* allergy to propofol, soy or peanuts
* history of central nervous system disease
* patient receiving a psychotropic treatment
* patient treated by a psychiatrist or a psychologist
* hypovolemia, high cardiovascular risk
* patients with a pace-maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Administered dose of propofol required to obtain the induction of anesthesia (bispectral index <60 for at least 30 seconds) | one hour

SECONDARY OUTCOMES:
calculated target plasma concentration corresponding to induction of anesthesia (bispectral index <60 for at least 30 seconds) | one hour
pain of injection | one hour
  Pain is assessed by two criteria:
  * withdrawal of the arm perfused (no = 0; withdrawal = 1; violent withdrawal = 2),
  * spontaneous expression (no = 0; frown = 1 grin = 2)
Hemodynamic consequences of induction of anesthesia | one hour
  Heart rate and blood pressure are measured just before induction of anesthesia and once it realized.
characteristics of the hypnotic procedure | one hour
  * For speed: focus obtained in a very fast (1), fast (2), medium (3), delayed (4), impossible to obtain (5).
  * For quality: very deep (1), deep (2), medium (3), superficial (4), not obtained (5)
Patient assessment of the induction of anesthesia | one hour
  4-point scale.
Time to loss of consciousness | one hour
  loss of eyelash reflex

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Szekely, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963